CLINICAL TRIAL: NCT01046786
Title: Safety and Feasibility of Umbilical Cord Blood Cell Transplant Into Injured Spinal Cord: an Open-Labeled, Dose-Escalating Clinical Tiral
Brief Title: Safety and Feasibility of Umbilical Cord Blood Cell Transplant Into Injured Spinal Cord
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: Chinese University of Hong Kong (Other); The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN102B
Record Dates: First submitted 2010-01-10; First posted 2010-01-12 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; cord blood mononuclear cell; Methylprednisolone; Lithium Carbonate
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Methylprednisolone; Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group A (Active Comparator): Intraspinal injection of 1.6 million cord blood mononuclear cell
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell
- Group B (Active Comparator): Intraspinal injection of 3.2 million cord blood mononuclear cell
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell
- Group C (Active Comparator): Intraspinal injection of 6.4 million cord blood mononuclear cell
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell
- Group D (Active Comparator): Intraspinal injection of 6.4 million cord blood mononuclear cell plus 30 mg/kg methylprednisolone
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell; Drug: Methylprednisolone
- Group E (Active Comparator): Intraspinal injection of 6.4 million cord blood mononuclear cell plus 30 mg/kg methylprednisolone plus 6 week course of oral lithium, titrated to maintain 0.6-1.0 mM serum level
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell; Drug: Methylprednisolone; Drug: Lithium

INTERVENTIONS:
Biological: Umbilical Cord Blood Mononuclear Cell — The cord blood mononuclear cells are obtained from thawed units of HLA-matched human umbilical cord blood. The cells will be slowly injected into the posterior gray matter after laminectomy and opening of the dura.
Drug: Methylprednisolone — 30 mg/kg methylprednisolone
  Arms: Group D; Group E
Drug: Lithium — oral lithium, titrated to maintain 0.6-1.0 mM serum level
  Arms: Group E

SUMMARY:
To investigate the feasibility, safety, efficacy and optimal dose of umbilical cord blood mononuclear cell transplant in the treatment of chronic spinal cord injuries.

DETAILED DESCRIPTION:
This is an open-label, dose-escalating clinical trial. Three groups of four patients will receive transplants of increasing doses of HLA-matched umbilical cord blood mononuclear cell into the spinal cord. In the fourth group, we will transplant the highest volume of cells that did not increase neurological deficits along with a single bolus of 30mg/kg methylprednisolone sodium succinate. In the fifth group of four subjects, we will inject that volume of cells plus a bolus intravenous dose of 30mg/kg methylprednisolone sodium succinate and a 6-week course of oral lithium carbonate titrated to 0.6-1.0 mM serum levels. All the subjects are encouraged to stand or walk for one hour a day after the cell transplantation.

The neurological and walking outcomes will be assessed 1, 2, 6, 24 and 48 weeks after transplantation. The outcomes of the five treatment groups will be compared by analysis of variance and, if possible, correlation with cell dose. Efficacy and safety will be analyzed comparing neurological change scores amongst the five different treatment groups. Loss of motor (>5 points) or sensor scores (>2 points) from baseline pre-treatment levels would be considered deleterious. Increases in scores above baseline would be considered beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender and 18-60 years old
* Subjects with chronic spinal cord injury (defined as ≧12 months post-initial SCI surgery) with stable neurological findings for at least 6 months
* Subject with a current neurological status of ASIA A
* The neurological level of the subjects is between C5 and T11
* The MRI shows that the injured site of the spinal cord is within three vertebral levels and there is no cyst
* Subjects must be able to read, understand, and complete the Visual Analog Scale
* Subjects who have voluntarily signed and dated an informed consent form, approved by the appropriate IRB, prior to any study-specific procedures

Exclusion Criteria:

* Significant renal, cardiovascular, hepatic and psychiatric diseases
* Significant medical diseases or infection (including but not limited to the carrier of hepatitis B virus or HIV)
* Pregnant or lactating woman
* Female of childbearing potential and who is unwilling to use an effective contraceptive method while enrolled in the study
* The MRI shows that the length of spinal cord lesion exceeds three segments or there is cyst in the spinal cord
* The lesion edge of the spinal cord cannot be determined by imaging technology
* Unavailability of HLA matched umbilical cord blood cells
* Any contraindication of laminectomy operation, MPSS and/or lithium carbonate
* Subject who is currently participating in another investigational study or has been taking any investigational drug within the last 4 weeks prior to screening of this study and finally
* Any criteria, which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol and/or would not be suitable to participant this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ASIA motor scores and sensory scores | 0, 1, 2, 6 24 and 48 weeks
ASIA Impairment Scale grade | 0, 1, 2, 6 24 and 48 weeks

SECONDARY OUTCOMES:
MRI and Diffusion Tensor Imaging of spinal cord | 0, 1, 24 and 48 weeks
Spinal Cord Independence Measure (SCIM) score | 0, 6, 24 and 48 weeks
Walking Index of Spinal Cord Injury (WISCI) level | 0, 6, 24 and 48 weeks
Modified Ashworth Scale (MAS) of Spasticity | 0, 1, 2, 6, 24 and 48 weeks
Visual Analog Scale (VAS) of pain | 0, 1, 2, 6, 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sang Poon, MD, Principal Investigator — The Chinese University of Hong Kong / Prince of Wales Hospital; Gilberto Leung, MD, Principal Investigator — The University of Hong Kong / Queen Mary Hospital
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin